CLINICAL TRIAL: NCT00967304
Title: REVERSEII: Validation of the "Men and HERDOO2"- A Clinical Decision Rule to Identify Patients With "Unprovoked" Venous Thromboembolism Who Can Discontinue Anticoagulants After 6 Months of Treatment.
Brief Title: Clinical Decision Rule Validation Study to Predict Low Recurrent Risk in Patients With Unprovoked Venous Thromboembolism
Acronym: REVERSEII
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: BioMérieux (Industry); Centre Hospitalier Régional et Universitaire de Brest (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2008039-01H
Record Dates: First submitted 2009-08-26; First posted 2009-08-27 (Estimated); Last update posted 2016-09-01 (Estimated); Status verified 2016-08

CONDITIONS: Idiopathic Venous Thromboembolism
Keywords: Unprovoked Venous thromboembolism; Clinical decision rule; Anticoagulants; Recurrence; Prognostic; Risk stratification
MeSH Terms: conditions — Recurrence | interventions — Clinical Decision Rules

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 Discontinue OAT or AAA (Experimental): Patients classified as being at low risk of recurrent VTE by the "HER DOO2"rule.
  If the clinical decision rule indicates that a patient is at low recurrence risk (<3% per year); anticoagulant therapy will be withdrawn and the participant will then be followed for 1 year for any VTE recurrence and/or bleeding.
  Interventions: Other: Application of the"Men continue and HER DOO2" rule
- 2 Observation arm (No Intervention): Men and patients classified as being at high risk of recurrent VTE by the "HER DOO2"rule.
  If the clinical decision rule indicates that a patient is at high recurrence risk then the decision to continue or discontinue anticoagulant therapy will be left to the discretion of physicians and patients as per current standard of care and this decision recorded. High risk patients (females classified as being at high risk of recurrent VTE by the CDR, and all males) will then be followed as an observational cohort for 1 year for any VTE recurrence and/or bleeding.

INTERVENTIONS:
Other: Application of the"Men continue and HER DOO2" rule — Consecutive patients will have the"Men continue and HER DOO2" rule applied by the attending physician between 5 - 12 months after treatment for a first unprovoked objectively proven major VTE.
  "Men continue and HER DOO2" rule: all men continue oral anticoagulants and women with 2 or more of the following features after 5-7 months of OAT should continue oral anticoagulants:1) HER - any Hyperpigmentation, Edema and Redness of either lower extremity, 2) Vidas D-dimer ≥250ug/L, 3) Obesity - BMI ≥30 kg/m2 and 4) Older age - Age ≥65 years.
  Other Names: Clinical Decision Rule
  Arms: 1 Discontinue OAT or AAA

SUMMARY:
The main objective of this study is to verify whether a new clinical decision rule identifying patients diagnosed with unprovoked blood clots who have a low risk of recurrence can safely stop oral anticoagulant therapy after 5-7 months of treatment.

DETAILED DESCRIPTION:
Up to 50% of patients with a first episode of venous thromboembolism (VTE) have no identifiable cause (i.e. are unprovoked VTEs). The risk of recurrent VTE in this large group of patients with unprovoked VTE after 3-6 months of anticoagulant therapy is 5-10.8% in the year following discontinuation of oral anticoagulant therapy. One in six to one in twenty recurrences of a new VTE are fatal. Given the intermediate risks of recurrence in unselected unprovoked VTE patients, clinicians do not have clear guidance on whether to continue or discontinue anticoagulants in patients with unprovoked VTE. Recently attention has turned to the concept of risk stratification to identify subgroups of patients with unprovoked VTE who could safely discontinue oral anticoagulation therapy (OAT).

In the REVERSE I study, a clinical decision rule derivation study conducted from 2001 to 2006, we developed and internally validated the clinical decision rule "Men continue and HER DOO2" that identifies patients with a first unprovoked VTE who likely have a low risk of recurrent VTE and could safely discontinue OAT subsequent to 5-7 months of OAT. The present study will evaluate if the "Men continue and HER DOO2" rule (comprised of gender, elevated D-dimer levels, post-thrombotic signs, obesity, and older age) is safe, clinically useful, and reproducible when prospectively implemented in multiple centers and a variety of settings. If this clinical decision rule is validated, it will provide physicians with important information to allow them to more confidently identify unprovoked VTE patients at low risk of VTE recurrence who may not need to continue OAT.

ELIGIBILITY:
Inclusion Criteria:

* First episode of major unprovoked VTE
* VTE objectively proven
* VTE treated for 5-12 months with anticoagulant therapy authorized for the REVERSE II study (initial or ongoing therapy)
* Absence of recurrent VTE during the treatment period

Exclusion Criteria:

* Less than 18 years of age
* Patients who have already discontinued anticoagulant therapy
* Patients requiring ongoing anticoagulation for reasons other than VTE
* Being treated for a recurrent unprovoked VTE
* Patients with high risk thrombophilia
* patients who plan on using exogenous estrogen(OCP,HRT)if anticoagulant therapy is discontinued
* Patients with pregnancy associated VTE
* Geographically inaccessible for follow-up
* Patients unable or unwilling to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2779 (Actual)
Dates: Start 2008-11; Primary Completion 2015-01 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
The primary study outcome is the incidence of adjudicated recurrent major VTE at 1 year in patients deemed by the "Men and HER DOO2" CDR to be at low risk of recurrent VTE. | One year

SECONDARY OUTCOMES:
Any VTE 1 year event rate in low risk patients | One year
Major bleeding 1 year event rate in un-anticoagulated low risk patients | One year
Major VTE 1 year event rate in high risk patients who continue anticoagulant therapy | One year
Major VTE 1 year event rate in high risk patients who discontinue anticoagulant therapy | One year
Major Bleeding 1 year event rate in high risk patients | One year
Clinical utility of the rule | One year
Inter-observer reliability of the clinical decision rule | One year

CONTACTS AND LOCATIONS:
Overall Officials: Marc Rodger, MD, MSc, Study Chair — Ottawa Hospital Research Institute
Locations (23):
- United States (3):
  - UC Davis, Santa Monica, California
  - Penobscot Bay Medical Center, Rockport, Maine
  - Duke University, Durham, North Carolina
- Prince of Wales Hospital, Sydney, New South Wales, Australia
- CUB Hopital Erasme, Brussels, Belgium
- Canada (12):
  - CDHA-Queen Elizabeth II Health Science Centre, Halifax, Nova Scotia
  - Hamilton Health Sciences Center, Hamilton, Ontario
  - Hamilton Health Sciences Corporation, Hamilton, Ontario
  - Victoria Hospital, London, Ontario
  - Ottawa Health Research Institute, Ottawa, Ontario
  - University Health Network, Toronto, Ontario
  - SMBD Jewish General Hospital, Montreal, Quebec
  - Hopital Sacre Coeur, Montreal, Quebec
  - McGill University Health Centre, Montreal, Quebec
  - St. Mary's Hospital - CHUM, Montreal, Quebec
  - Hopital Enfant Jesus, Québec, Quebec
  - Saskatchewan Drug Research Institute, Saskatoon, Saskatchewan
- Centre Hospitalier Regional Universitaire de Brest, Brest, France
- India (4):
  - Orange Lifesciences, Nirmaya
  - Sahyadri Speciality Hospital, Pune
  - Shefali Centre, Shefali
  - Jashvant Patel Clinic, Surat
- Hopitaux Universitaires de Geneve, Geneva, Switzerland

REFERENCES:
- [Background] Rodger MA, Kahn SR, Wells PS, Anderson DA, Chagnon I, Le Gal G, Solymoss S, Crowther M, Perrier A, White R, Vickars L, Ramsay T, Betancourt MT, Kovacs MJ. Identifying unprovoked thromboembolism patients at low risk for recurrence who can discontinue anticoagulant therapy. CMAJ. 2008 Aug 26;179(5):417-26. doi: 10.1503/cmaj.080493. PMID 18725614
- [Derived] Rodger MA, Le Gal G, Anderson DR, Schmidt J, Pernod G, Kahn SR, Righini M, Mismetti P, Kearon C, Meyer G, Elias A, Ramsay T, Ortel TL, Huisman MV, Kovacs MJ; REVERSE II Study Investigators. Validating the HERDOO2 rule to guide treatment duration for women with unprovoked venous thrombosis: multinational prospective cohort management study. BMJ. 2017 Mar 17;356:j1065. doi: 10.1136/bmj.j1065. PMID 28314711